CLINICAL TRIAL: NCT06357481
Title: Evaluation of Postoperative Pain After Single Visit Retreatment of Symptomatic and Asymptomatic Teeth With Minimal Invasive Rotary and Reciprocal Nickel Titanium Files: A Randomized Clinical Trial
Brief Title: Evaluation of Postoperative Pain After Single Visit Retreatment of Symptomatic and Asymptomatic Teeth
Acronym: Endodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SaglikBilimleriU-22-122
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Post-operative Pain; Retreatment; Symptomatic Periapical Periodontitis; Endodontic Disease; Asymptomatic Periapical Periodontitis
Keywords: Post-operative pain; Minimal invasive files; Single visit; Retreatment; Remover files
MeSH Terms: conditions — Pain, Postoperative; Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: Eighty patients who needed endodontic retreatment were assingned to 2 groups according to symptomatic or asymptomatic teeth and 4 subgroups with rotary and resiprocal files.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MICRO MEGA ONE RECI FILES in Group 1 (Experimental): During the non-surgical retreatments, the rotary file systems used in our treatment consist of One Reci system 25.04, 25.06, 35.04, and 45.04 files in symptomatic teeth.
  Interventions: Procedure: Endodontic Retreatment
- MICRO MEGA ONE CURVE MINI FILES in Group 2 (Experimental): During the non-surgical retreatments, the rotary file systems used in our treatment consist of One Curve mini system 25.04, 25.06, 35.04, and 45.04 files in symptomatic teeth.
  Interventions: Procedure: Endodontic Retreatment
- MICRO MEGA ONE RECI FILES in Group 3 (Experimental): During the non-surgical retreatments, the rotary file systems used in our treatment consist of One Reci system 25.04, 25.06, 35.04, and 45.04 files in asymptomatic teeth.
  Interventions: Procedure: Endodontic Retreatment
- MICRO MEGA ONE CURVE MINI FILES in Group 4 (Experimental): During the non-surgical retreatments, the rotary file systems used in our treatment consist of One Curve mini system 25.04, 25.06, 35.04, and 45.04 files in asymptomatic teeth.
  Interventions: Procedure: Endodontic Retreatment

INTERVENTIONS:
Procedure: Endodontic Retreatment — A single operator procedured in one visit of non-surgical endodontic retreatment. Teeth were anesthetized using articaine hydrochloride with epinephrine 1:200,000 for mandibulary premolar teeth with one root canal. Each tooth was isolated with a rubber dam and then coronal restorations and caries were removed using sterile high-speed burs under water cooling. After preperation of the cavity access and localization of the canal orifice, all microorganisms that may have entered the root canal system are eliminated by removing the old canal filling with the One Flare and MicroMega REMOVER files in the MicroMega retreatment kit.

SUMMARY:
Introduction: The aim of this study comparing the post operative pain after the retreatment of asymptomatic and symptomatic teeth that during single visit treatment with rotary and reciprocal nickel titanium files.

Methods: One hundred and forty one patients scheduled for non-surgical endodontic retreatment were included for evaluation. Eighty five patients who needed endodontic retreatment were assingned to 2 groups according to semptomatic or asemptomatic teeth and 4 subgroups with rotary and resiprocal files. Endodontic filling material was removed with One Flare and MicroMega REMOVER files in the retreatment kit. Patients then recorded their postoperative pain on a VAS scale at 24h, 48h, 72h, 7 days and 14 days post-treatment. Results were analyzed using the Shapiro-Wilk, Mann-Whitney U, Kruskal-Wallis, Dunn-Bonferroni and Pearson Chi-square tests.

DETAILED DESCRIPTION:
Retreatment is the procedure performed to regain healthy periapical tissues that the teeth have undergone root canal treatment are re-infected due to apical or coronal leakage, or after an inadequate root canal treatment. When primary root canal treatment fails, the first treatment option is non-surgical retreatment to eliminate the infection. In general, the reported success rate of retreatment ranges from 62% to 91%.

This randomized clinical study's primary goal is to evaluate the postoperative pain following a single visit of root canal retreatment for asymptomatic and symptomatic mandibular premolars using reciprocal and rotary file systems. Therefore, this study aims to compare the effect of one curve mini (rotary file system) and one reci (resiprocal file system) nickel-titanium file systems on postoperative pain after non surgical endodontic retreatment within symptomatic and asymptomatic teeth.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Apical Periodontitis
* Asymptomatic Apical Periodontitis
* Adult patients between 18-67 years aged

Exclusion Criteria:

* Patient under 18 years old
* Complicating systemic disease
* Allergies to local anesthetic agents
* Acute apical abscesses
* Periodontal pockets deeper than 5 mm or more mobilty than level 1
* Bruxist and teeth-grinding patient
* Pregnant women
* Presence of external root resorption
* Root fracture
* Root perforation
* Calcified root canals

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | Day 1, Day 2, Day 3, Day 7 and Day 14
  After repeated root canal treatments, postoperative pain is frequent. The response to pain varies depending on the situation and perception of pain is not always continuous. The pain was evaluated with a visual analog scale (VAS) (0: no pain, 1-2: discomfort, 3-4: mild, 5: moderate, 6-7: severe, 8-9: very severe, 10: worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Gurkan Gunec, Asst Prof, Study Director — Saglik Bilimleri University
Locations (1):
- Hüseyin Gürkan Güneç, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only after the results of the study are published in one of the international journals, they can be made available for the benefit of researchers, while any other data will not be shared.

REFERENCES:
- [Result] Nagendrababu V, Duncan HF, Bjorndal L, Kvist T, Priya E, Jayaraman J, Pulikkotil SJ, Dummer PMH. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: explanation and elaboration. Int Endod J. 2020 Jun;53(6):774-803. doi: 10.1111/iej.13304. Epub 2020 May 9. PMID 32266988
- [Derived] Gunec HG, Pehlivan B, Topbas C, Kul AK, Sirin DA. Postoperative Pain Following Single-Visit Nonsurgical Retreatment Using Minimally Invasive Rotary vs. Reciprocating Nickel-Titanium File Systems: A Two-Arm Parallel Randomized Clinical Trial. Pain Res Manag. 2025 Sep 8;2025:6826535. doi: 10.1155/prm/6826535. eCollection 2025. PMID 40958962
- See also: Guidelines for reporting randomized trials in Endodontics — https://pubmed.ncbi.nlm.nih.gov/32266988/
- Available data/document: Study Protocol: doi: 10.1111/iej.13304 — https://pubmed.ncbi.nlm.nih.gov/32266988/